CLINICAL TRIAL: NCT01769521
Title: A Single Center, Prospective, Open Label Study Assessing the Relationship Between the 24-hour Intraocular Pressure Pattern as Determined by Sensimed Triggerfish® and the 24-hour Blood Pressure Pattern in Patients With Primary Open Angle Glaucoma
Brief Title: Relationship Between 24-hour IOP Pattern and the 24-hour Blood Pressure Pattern in Patients With POAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TF-1011
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Primary Open Angle Glaucoma; Normal Tension Glaucoma
Keywords: Glaucoma; IOP; Blood pressure; ECG
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triggerfish (Experimental): Device: Sensimed Triggerfish
  Interventions: Device: Sensimed Triggerfish®

INTERVENTIONS:
Device: Sensimed Triggerfish® — Portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours

SUMMARY:
Interplay between the increasing IOP and decreasing blood pressure (BP) during the 24-hour period, especially in the nocturnal period, may lead to insufficient perfusion pressure of the optic nerve and contribute to the glaucomatous damage in adjunct to the antero-posterior vectorial mechanical impact on the lamina cribrosa, the translaminar pressure. Patients with progressive VF loss showed greater nocturnal BP dips than patients with stable VF. Reduced mean intraocular perfusion pressure (IOPP) was significantly associated with the extent of glaucomatous damage. How the nycthemeral IOP fluctuation influences glaucoma progression has not been studied in a prospective manner and remains to be elucidated.

The purpose of this study is to assess the relationship between the 24-hour IOP fluctuation pattern and the 24-hour BP pattern in patients with primary open angle glaucoma (POAG). IOP fluctuations will be monitored with SENSIMED Triggerfish®, a portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG, including progressing normal tension glaucoma (NTG) based on recent or recurrent disc haemorrhage
* No anti-glaucomatous drug treatment or washed-out for a period of 4 weeks prior to SD0 and absent throughout the study
* Aged more than 18 years, of either sex
* Not more than 4 diopters spherical equivalent on both eyes
* Not more than 2 diopters cylinder equivalent on both eyes
* Have given written informed consent, prior to pre-study screening

Exclusion Criteria:

* Patients with history of ocular surgery within the last 3 months
* Corneal or conjunctival abnormality hindering contact lens adaptation
* Severe dry eye
* Secondary forms of OAG
* Patients with systemic hypertension
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Wear of full frame metallic glasses during Triggerfish® monitoring
* Patients not able to understand the character and individual consequences of the investigation
* Simultaneous participation in other clinical research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between the 24-hour IOP fluctuations as monitored by Triggerfish® and the 24-hour blood pressure pattern in patients with POAG. | 24-hour

SECONDARY OUTCOMES:
Nycthemeral IOP pattern | 24-hour
  The nycthemeral IOP fluctuation pattern, will be derived from the Triggerfish®, over a 24-hour period. Curves will be plotted for the IOP fluctuation.
Relationship between the nocturnal IOP fluctuation pattern and the diurnal fluctuation pattern (office hours) | 24 hours
  The nocturnal IOP fluctuation pattern will be compared to that of the diurnal fluctuation pattern (office hours). The diurnal IOP fluctuation pattern will be compared to the tonometric IOP curve concomitantly assessed in the contralateral eye.
Relationship between intraocular pulsation amplitude and BP | 24-hours
  The relationship between intraocular pulsation amplitude and BP will be determined by the determination of the mean intraocular Triggerfish output (IOT), SIOT and DIOT and correlated to the mean BP, SBP and DBP.
Relationship between the intraocular pulsation frequency and heart rate (HR) | 24-hours
  The relationship between the intraocular pulsation frequency as determined by Triggerfish® will be correlated with the heart frequency as determined by ECG
Assess safety and tolerability | 24-hours
  AEs and SAEs will be collected throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Kocięcki, MD, Principal Investigator — Przemienienia Pańskiego Hospital
Locations (1):
- Przemienienia Pańskiego Hospital, Poznan University of Medical Sciences Karol Marcinkowski, Poznan, Poland